CLINICAL TRIAL: NCT05829148
Title: Comparison Between the Effect of Dexmedetomidine, Melatonin and Pregabalin on Hypotensive Anesthesia in Patients Undergoing Functional Endoscopic Sinus Surgery
Brief Title: The Effect of Dexmedetomidine, Melatonin and Pregabalin
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Alaa Abdel-Khalek
Record Dates: First submitted 2023-04-08; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Endoscopic Sinus Surgery
MeSH Terms: interventions — Dexmedetomidine; Melatonin; Pregabalin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dexmedetomidine Group (Active Comparator): This Group about 30 patients will receive dexmedetomidine loading dose 1 µg/kg over a period of 15 minutes and maintenance 0.2µg/kg/h throughout the surgery .
  Interventions: Drug: Dexmedetomidine
- Melatonin Group (Active Comparator): This Group about 30 patients will receive 10 mg melatonin (2 tablets) one hour before starting of the operation.
  Interventions: Drug: Melatonin
- Pregabalin Group (Active Comparator): This Group about 30 patients will receive oral pregabalin 150 mg one hour before starting of the operation..
  Interventions: Drug: Pregabalin
- Control Group (Placebo Comparator): This Group about 30 patients will receive oral starch tablet as a control. Heart rate (HR) and blood pressure values will be recorded at various intervals.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Comparison the effect of Dexmedetomidine, Melatonin and Pregabalin on hemodynamics, recovery profile and postoperative pain in patients undergoing Functional endoscopic sinus
  Arms: Dexmedetomidine Group
Drug: Melatonin — Melatonin
  Arms: Melatonin Group
Drug: Pregabalin — Pregabalin
  Arms: Pregabalin Group
Drug: Placebo — Placebo
  Arms: Control Group

SUMMARY:
Various drugs have been used for the purpose: nitroglycerine, sodium nitroprusside, propofol, beta blockers, calcium channel blockers, higher concentrations of inhalational anesthetics etc. Since all these drugs have certain limitations there was a search for more safe and effective drug

DETAILED DESCRIPTION:
Functional Endoscopic Sinus Surgery (FESS) is done via endoscope and the area is highly vascular thus it becomes important to minimize bleeding, hence we require hypotensive anesthesia.

Dexmedetomidine (a highly selective α2-receptor agonist that has sedative, analgesic, anxiolytic, and opioid sparing effects without significant respiratory depression) it also reduces the need for inhaled anesthetics. dexmedetomidine also minimizes postoperative opioid consumption as well as nausea, vomiting, and anxiety.

Melatonin is a neurohormone mainly secreted from the pineal gland by the suprachiasmatic nucleus. It possesses a circadian secretion pattern and regulates the biological clock; it also offers antiemetic, analgesic, and anxiolytic effects. Due to its effect on both acute and chronic pain, melatonin (available in 5mg tablet form) fulfills a beneficial role in reducing postoperative opioid consumption while minimizing nausea and vomiting.

Pregabalin, whose structure is similar to the inhibitory neurotransmitter gamma-aminobutyric acid (GABA), possesses analgesic and anxiolytic activities and is effective in alleviating the neuropathic component of acute nociceptive pain of surgery. It has also been used as premedication to attenuate the hemodynamic stress response to laryngoscopy and intubation and to decrease intraoperative anesthetic requirement

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing Functional endoscopic sinus surgery (ASA I & II)

Exclusion Criteria:

- Hepatic, renal, endocrinal, hematological disorders.

* BMI>30 kg/m2.
* Patients receiving magnesium supplementation, anticonvulsant drugs or antipsychotic drugs.
* Chronic use of opioids.
* Current treatment with β-blocker or calcium channel blocker.
* Known allergies to any of study drugs.
* Patients refusal to the study

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Pain Relieve | 2 hours post operative
  Assessment of the pain post-operatively in patients with pain score by VAS as : Total scores vary from 0 to 10 in this method, with a higher score indicating more severe pain,

SECONDARY OUTCOMES:
controlled pulse rate | From base line to 1 hour after the end of the operation
  Hemodynamics stability
controlled blood pressure | From base line to 1 hour after the end of the operation
  Hemodynamics stability

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AbdelGawad, Assist.Prof, Study Chair — Al-Azhar University, Faculty of medicine for boys
Locations (1):
- Al-Azhar University hospitals, Cairo, Egypt